CLINICAL TRIAL: NCT07007598
Title: Prevention of Post-Polypectomy Colorectal Bleeding by Clips in Patients on Anticoagulants: a Retrospective Single Center Propensity Score Analysis
Brief Title: Prevention of Post-Polypectomy Colorectal Bleeding by Clips in Patients on Anticoagulants
Acronym: PiCAnt
Status: Recruiting | Type: Observational
Sponsor: Helios Kliniken Schwerin (Other)
Collaborators: Medical School Hamburg (Other)
Responsible Party: Principal Investigator, Dr. med. Daniel Schmitz, Head Physician, Helios Kliniken Schwerin
Other Study IDs: HeliosSchwerin GAS 01
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Polyp of Colon
Keywords: polyps; Hemorrhage; Anticoagulants
MeSH Terms: conditions — Colonic Polyps; Polyps; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal polypectomy and prophylactic clipping before restarted anticoagulants: At least one prophylactic clip is applied to close the mucosal defect after polypectomy
  Interventions: Device: Hemostatic clip
- Colorectal polypectomy without prophylactic clipping before restarted anticoagulant: A prophylactic clip is not applied to close the mucosal defect after polypectomy.

INTERVENTIONS:
Device: Hemostatic clip — The hemostatic clip is endoscopically applied after a colorectal polypectomy to close the mucosal defect.
  Groups: Colorectal polypectomy and prophylactic clipping before restarted anticoagulants

SUMMARY:
This observational study aims to retrospectively determine if clips can prevent post-polypectomy bleeding in adults who have received restarted anticoagulants after a colorectal polypectomy, using a large, single-center patient registry.

The main question it aims to answer is:

Can clips prevent post-polypectomy bleeding in adults who have received restarted anticoagulants after a colorectal polypectomy? Researchers will compare adults who received preventive clipping after a polypectomy with those who did not, regarding colorectal bleeding after receiving restarted anticoagulants.

Participants have undergone a colorectal polypectomy and received restarted anticoagulants (acetylsalicylic acid excluded) after the procedure.

DETAILED DESCRIPTION:
Screening colonoscopy allows early detection of cancer and removal of adenomas before they become malignant. Unresected polyps larger than 1 cm have a 24% risk of invasive adenocarcinoma. Post-polypectomy bleeding is influenced by factors such as polyp size, location, tumor type, anticoagulants and concomitant diseases. Prophylactic measures such as clipping show mixed results; selective clipping is cost-effective, but universal clipping is not. The updated ESGE guideline on colorectal polypectomy and endoscopic mucosal resection from 2024 recommends prophylactic endoscopic clip of the mucosal defect after endoscopic mucosal resection of large non-pedunculated polyps in the right colon to reduce the risk of delayed bleeding. However, there is no clear recommendation for patients on anticoagulants whether to use or not to use prophylactic clipping. Therefore, this observational study aims to retrospectively determine if clips can prevent post-polypectomy bleeding in adults who have received restarted anticoagulants after a colorectal polypectomy, using a large, single-center patient registry (> 10.000 colonoscopies).

ELIGIBILITY:
Inclusion Criteria:

* adult who has received a colonoscopy with endoscopic colorectal polypectomy
* patient who has received at least one anticoagulant after polypectomy

Exclusion Criteria:

* Endoscopic polypectomy was combined with closure of the mucosal defect by a suturing device or full thickness resection device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have received an endoscopic colorectal polypectomy
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Colorectal Post-polypectomy bleeding | Up to 30 days after colorectal endoscopic polypectomy
  Mucosal defect-associated bleeding after removal of a colorectal polyp bei endoscopic polypectomy.
  The metachronous interval bleeding rate is calculated by dividing the number of bleeding events by the number of colonoscopies with polypectomy. The following are counted as polypectomy bleeding:
  1. Polypectomy bleeding is visualized directly during a subsequent colonoscopy.
  2. Polypectomy bleeding is considered probable if a subsequent colonoscopy is performed due to lower gastrointestinal bleeding, and evidence of blood is found in association with the polypectomy.
  3. Polypectomy bleeding is considered probable if the patient was hospitalized for monitoring or had his hospital stay extended because he showed visible perianal bleeding. However, a colonoscopy was not performed because the bleeding had stopped spontaneously and/or the risk of a subsequent colonoscopy was deemed too high in relation to the potential benefits.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Schmitz, Dr.med., Principal Investigator — Helios Kliniken Schwerin
Locations (1):
- Helios Kliniken Schwerin, Schwerin, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Nishad N, Thoufeeq MH. Post-polypectomy colorectal bleeding: current strategies and the way forward. Clin Endosc. 2025 Mar;58(2):191-200. doi: 10.5946/ce.2024.241. Epub 2024 Nov 27. PMID 39722137
- [Background] Ferlitsch M, Hassan C, Bisschops R, Bhandari P, Dinis-Ribeiro M, Risio M, Paspatis GA, Moss A, Libanio D, Lorenzo-Zuniga V, Voiosu AM, Rutter MD, Pellise M, Moons LMG, Probst A, Awadie H, Amato A, Takeuchi Y, Repici A, Rahmi G, Koecklin HU, Albeniz E, Rockenbauer LM, Waldmann E, Messmann H, Triantafyllou K, Jover R, Gralnek IM, Dekker E, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2024. Endoscopy. 2024 Jul;56(7):516-545. doi: 10.1055/a-2304-3219. Epub 2024 Apr 26. PMID 38670139